CLINICAL TRIAL: NCT05139979
Title: Yogic Breathing and Guided Meditation for Long Covid Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021P000552
Record Dates: First submitted 2021-09-23; First posted 2021-12-01 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Stress; Shortness of Breath
Keywords: Long COVID-19; Mental health; Anxiety; Stress; Breathing; Meditation; Yoga; Isha Kriya
MeSH Terms: conditions — COVID-19; Dyspnea; Post-Acute COVID-19 Syndrome; Psychological Well-Being; Anxiety Disorders; Respiratory Aspiration | interventions — Respiration

STUDY DESIGN:
Intervention Model Description: Upon enrollment and randomization, the intervention group will be followed weekly for 3 weeks as well as on week 6. The waitlisted control group will be followed for 3 weeks as controls and will then learn the intervention and be followed for additional 3 weeks (total of 6 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Webinar-Based Intervention (Experimental): Breathing and Wellness Webinar: two yogic breathing practices (Simha Kriya and Naddi Shuddi) and a guided meditation (Isha Kriya).
  Interventions: Behavioral: Breathing and Wellness Webinar
- Control (Placebo Comparator): This group will be asked to wait for 3 weeks before being introduced to the Breathing and Wellness Webinar intervention which includes two yogic breathing practices (Simha Kriya and Naddi Shuddi) and a guided meditation (Isha Kriya).
  Interventions: Other: Routine Daily Activity

INTERVENTIONS:
Behavioral: Breathing and Wellness Webinar — Simha Kriya : a 3-minute energizing breathing practice to expand lung capacity and improve immunity, to be practiced twice daily.
  Nadi Shuddhi - a gentle 4-minute breathing practice for creating mental balance and relaxation, to be practiced for a minimum of 4 minutes daily.
  Isha Kriya - a 15-minute guided meditation that incorporates the breath and the awareness to create mental clarity and health, to be practiced at least once (ideally twice) daily.
  Arms: Webinar-Based Intervention
Other: Routine Daily Activity — Participants in the control group are asked to perform routine daily activities until enrolled into the intervention arm.
  Arms: Control

SUMMARY:
This study aims to assess the impact of brief digitally delivered breathing practice and guided meditation on post-Covid physical and mental symptoms in Long Covid Patients.

DETAILED DESCRIPTION:
Long Covid symptoms can last weeks to months after the initial Covid infection or can appear weeks after. It can occur in those with mild disease or asymptomatic patients. Most commonly reported symptoms of Long Covid are:

* Tiredness or fatigue
* Difficulty thinking or concentrating (sometimes referred to as "brain fog")
* Headache
* Loss of smell or taste
* Dizziness on standing
* Fast-beating or pounding heart (also known as heart palpitations)
* Chest pain
* Difficulty breathing or shortness of breath
* Cough
* Joint or muscle pain
* Depression or anxiety
* Fever
* Symptoms that get worse after physical or mental activities

To this date, nearly 180 million people have been infected with Covid19 and over 3 million have lost their lives worldwide. The increasing prevalence of patients with Long Covid symptoms and the lack of effective solutions to address their condition, creates an urgent need for non-pharmacological interventions that are effective and scalable and can be delivered online to accommodate for the limitations due to the Covid pandemic.

Yogic Breathing and Meditation techniques have been shown to have various health benefits including improving pulmonary function and mental health. Prominent health institutions are recommending breathing exercise to their Covid patients to assist their respiratory recovery9. Meditation and breathing is also shown to help with Covid related stress and anxiety.

This study is a waitlisted randomized controlled trial conducted in 2 phases:

Phase 1: If participants are in the intervention group, they will be asked to learn and practices two Yogic Breathing practices (Simha Kriya and Nadi Shuddhi) and a guided meditation (Isha Kriya) for 3 weeks They will be asked to complete a set of questionnaires at baseline and the end of each week. Participants in the waitlisted control group will be asked to perform their regular daily routine as they wait to be enrolled into the intervention at the end of 3 weeks. The waitlisted control group will also be recruited for semi-structured individual interviews during this time.

Phase 2: The waitlisted control group will begin the intervention at week 3 and continue until week 6. They will be asked to continue completing the questionnaires at the end of each week. The intervention group will be asked to complete a final follow-up questionnaire at the end of week 6. The intervention group will also be recruited for semi-structured individual interviews during this time.

Focus group discussions with both the intervention and control groups are conducted at the end of the study to collect general information about the participant's general experience with the current study and what matters to them as a Long COVID patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Interested in attending the online Breathing and Wellness webinar.
* Laboratory-confirmed (PCR) history of Covid-19 infection.
* Long Covid condition diagnosis by a physician.
* Able to read and comprehend English.
* Currently residing in the United States.

Exclusion Criteria:

● Any medically limiting diagnosis that prevents a patient from doing the intervention or completing the assessments as determined by the PI such as severe Major Depression (under medication), Schizophrenia, Bipolar disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Compliance | For Phase 1 analysis: Baseline to 3 weeks. For Phase 2 analysis: Baseline to 6 weeks.
  The weekly compliance questionnaire is a tool which helps the participants to keep track of their activities each week. This enables the study team to measure compliance and protocol adherence by the participants by collecting information on their routine activity practiced and its frequency. This will be reported in "Number of days an intervention was practiced in a week". Compliance is defined as completing 60% (4 days/week or more) of the activity that is prescribed in the protocol. This means that at least one of the three practices (Isha Kriya, Nadi Shuddhi, or Simha Kriya) must be completed once a day for a minimum of four days.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | For Phase 1 analysis: Baseline to 3 weeks. For Phase 2 analysis: Baseline to 6 weeks.
  PSS is a 10-question validated instrument that assesses stress. Participants are asked to rate on a scale of 0 (never) to 4 (very often) how often they agree with various statements.
Profile of Mood States (POMS) | For Phase 1 analysis: Baseline to 3 weeks. For Phase 2 analysis: Baseline to 6 weeks.
  This is a short validated survey used to measure six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A five-point scale ranging from "not at all" to "extremely" is administered and scores for each dimension contributes to calculation of positive and negative subscales in conjunction to total mood disturbance.
Quality of Life Survey (SF12) | For Phase 1 analysis: Baseline to 3 weeks. For Phase 2 analysis: Baseline to 6 weeks.
  SF12 is a validated self-reported measure of the impact of health on everyday quality of life. It evaluates domains of physical activities, social activities, usual role activities, bodily pain, general mental health, vitality and general health perception.
Multidimensional Dyspnea Profile (MDP) | For Phase 1 analysis: Baseline to 3 weeks. For Phase 2 analysis: Baseline to 6 weeks.
  MDP is a validated scale to assess the overall breathing discomfort, sensory qualities and emotional responses using 8 questions. It is not intended for a particular activity and can be used during rest, activity or during clinical care. For assessing Long Covid patients, the first three parts (breathing discomfort and sensory qualities) are commonly used.
Somatic Symptom Scale 8 Items (SS8) | For Phase 1 analysis: Baseline to 3 weeks. For Phase 2 analysis: Baseline to 6 weeks.
  SS8 is a validated brief questionnaire to assess common somatic symptoms including pain, shortness of breath, dizziness, fatigue and trouble sleeping. Participants are asked to rate on a scale of 0 (not at all) to 4 (very much) how often they agree with various statements. Items from each of the 8 questions are then summed to create a total perceived stress score.
Qualitative Assessments | For Phase 1 analysis: Baseline to 3 weeks. For Phase 2 analysis: Baseline to 6 weeks.
  The semi-structured individual interviews will allow us to gain rich, descriptive information about the participant's experience with the long COVID symptoms, treating physicians, and the effect of the provided practices on their symptoms. The focus group interviews will be semi-structured to ensure a systematic and flexible approach to data collection, allowing us to gain rich information about the participant's general experience with the current study and what matters to them as a Long COVID patients.
  The interviews will cover the following main topics: (1) Perceptions of the participants on their long COVID symptoms, (2) Perceptions of the participants on their treating physicians (3) the effect of the provided meditation practices on their long COVID symptoms (4) and what matters to the Long COVID patients as well as their general experience as participants in the current study.

CONTACTS AND LOCATIONS:
Overall Officials: Balachundar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

REFERENCES:
- [Background] Greenhalgh T, Knight M, A'Court C, Buxton M, Husain L. Management of post-acute covid-19 in primary care. BMJ. 2020 Aug 11;370:m3026. doi: 10.1136/bmj.m3026. No abstract available. PMID 32784198
- [Background] Taquet M, Geddes JR, Husain M, Luciano S, Harrison PJ. 6-month neurological and psychiatric outcomes in 236 379 survivors of COVID-19: a retrospective cohort study using electronic health records. Lancet Psychiatry. 2021 May;8(5):416-427. doi: 10.1016/S2215-0366(21)00084-5. Epub 2021 Apr 6. PMID 33836148
- [Background] Abel AN, Lloyd LK, Williams JS. The effects of regular yoga practice on pulmonary function in healthy individuals: a literature review. J Altern Complement Med. 2013 Mar;19(3):185-90. doi: 10.1089/acm.2011.0516. Epub 2012 Sep 14. PMID 22978245
- [Background] Budhi RB, Payghan S, Deepeshwar S. Changes in Lung Function Measures Following Bhastrika Pranayama (Bellows Breath) and Running in Healthy Individuals. Int J Yoga. 2019 Sep-Dec;12(3):233-239. doi: 10.4103/ijoy.IJOY_43_18. PMID 31543632
- [Background] Rangasamy V, Thampi Susheela A, Mueller A, F H Chang T, Sadhasivam S, Subramaniam B. The effect of a one-time 15-minute guided meditation (Isha Kriya) on stress and mood disturbances among operating room professionals: a prospective interventional pilot study. F1000Res. 2019 Mar 26;8:335. doi: 10.12688/f1000research.18446.1. eCollection 2019. PMID 32665843
- [Background] Maric V, Mishra J, Ramanathan DS. Using Mind-Body Medicine to Reduce the Long-Term Health Impacts of COVID-Specific Chronic Stress. Front Psychiatry. 2021 Feb 22;12:585952. doi: 10.3389/fpsyt.2021.585952. eCollection 2021. No abstract available. PMID 33692706
- [Background] Rain M, Subramaniam B, Avti P, Mahajan P, Anand A. Can Yogic Breathing Techniques Like Simha Kriya and Isha Kriya Regulate COVID-19-Related Stress? Front Psychol. 2021 Apr 15;12:635816. doi: 10.3389/fpsyg.2021.635816. eCollection 2021. PMID 33935886
- [Background] Narayanan S, Tennison J, Cohen L, Urso C, Subramaniam B, Bruera E. Yoga-Based Breathing Techniques for Health Care Workers During COVID-19 Pandemic: Interests, Feasibility, and Acceptance. J Altern Complement Med. 2021 Aug;27(8):706-709. doi: 10.1089/acm.2020.0536. Epub 2021 Apr 9. PMID 33835830
- See also: Related Info — http://www.mayoclinic.org/diseases-conditions/coronavirus/in-depth/coronavirus-long-term-effects/art-20490351
- See also: Related Info — http://covid19.who.int
- See also: Related Info — http://www.hopkinsmedicine.org/health/conditions-and-diseases/coronavirus/coronavirus-recovery-breathing-exercises